CLINICAL TRIAL: NCT02756234
Title: Implementing Myocardial Computed Tomographic Perfusion in a Community Hospital Setting
Status: Completed | Type: Observational
Sponsor: Lancaster General Hospital (Other)
Collaborators: Toshiba America Medical Systems, Inc. (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-9-LGH
Record Dates: First submitted 2016-04-22; First posted 2016-04-29 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Qualifying CTP patients: A convenience sample of all qualifying patients for CTP procedure

SUMMARY:
The objective of this study is to carefully monitor all patients undergoing Computed Tomographic Perfusion (CTP) at Lancaster General Hospital for safety, and determine the efficiency of the CTP procedure in a community setting.

DETAILED DESCRIPTION:
This will be a prospective, observational study designed to include a convenience sample of all qualifying patients undergoing myocardial CTP.

The study will enroll patients who have undergone a clinically indicated CCTA for suspicion of coronary artery disease and have a suspected coronary stenosis ≥50%-69% on that examination. CCTA is a clinically indicated and standard of care procedure at Lancaster General Hospital. This pilot study will enroll a convenience sample of fifteen (15) patients at Lancaster General Hospital who satisfy all study criteria.

When a patient has a coronary CTA, physician co-investigators, all of whom are certified by the Certification Board of Cardiovascular Computed Tomography and credentialed by Johns Hopkins for CTP, will evaluate the scan for the presence of lesions that would qualify the patient for inclusion. Patients with lesions between 50% and 70% will be approached for participation in the CTP study(37). Those who agree to participate will be scheduled to have the CTP performed within thirty (30) days of the initial Coronary CTA procedure.

The CTP procedure involves infusion of a stress agent and a contrast bolus prior to image acquisition. The CTP examination will be graded using the standard 17-segment myocardial model recommended by the ACCF/AHA for nuclear myocardial perfusion and stress echocardiography, in comparison to the myocardial appearance from the baseline coronary CTA. Areas of myocardial hypo-enhancement (decreased CT signal) under hyperemic conditions (coronary vasodilation during the regadenoson infusion) indicate possible ischemia.

If a coronary stenosis is severe enough to reduce myocardial perfusion, then studies have shown that an invasive therapy that includes revascularization offers benefit to the patient. Use of CTP may allow the investigators to determine, with improved accuracy, if patients have hemodynamically significant coronary stenoses. These results will be reported to the patients' treating physicians and may be used in treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Index CCTA. The patient must have a CCTA done for clinical indications within the 2 weeks prior to consent/enrollment, ordered by The Heart Group of Lancaster General Health.
* Age greater than 18 years.
* Lesion(s) requiring further testing. Upon review of the coronary CT angiogram, the interpreting physician (who was trained at the Johns Hopkins course for CTP imaging) finds at least one lesion that could benefit from further evaluation, specifically at least one stenosis of 50%-70%, or lesions with unclear stenosis severity suspected of being 50%-70%.
* Referring physician agreement. The referring physician has been contacted and agrees that the patient can be approached for consent.
* Informed consent. The patient is willing and able to provide informed consent.

Exclusion Criteria:

* CCTA complication. After an observation period of at least 20 minutes after the index CCTA, any evidence of MACE, allergy, or any other untoward clinical event that reduces CTP safety or suitability (as defined by attending physician) will exclude a patient from eligibility.
* Contraindication to regadenosen according to LGH protocol (addendum 2).
* Medical record of acute ischemia as evidenced on ECG or positive cardiac biomarkers in the interim between CCTA and CTP. Electrocardiographic evidence of acute ischemia includes acute STEMI (ST elevation equal to or greater than 1mm in two or more leads), ST segment depression and/or T wave inversion (not known to be old and thought to be evidence of ongoing ischemia). Positive cardiac biomarkers include elevated troponin, myoglobin, and/or creatinine phosphokinase MB fraction).
* History of asthma or chronic obstructive pulmonary disease requiring bronchodilators or steroid therapy within the past 3 months.
* Inability to tolerate beta blockers.
* Atrio-ventricular block (Type II-III), prolonged QT interval or sick sinus syndrome.
* Renal insufficiency (creatinine ≥1.6 and/or, GFR < 60 ml/m) or renal failure requiring dialysis.
* Atrial fibrillation or other markedly irregular rhythm.
* Psychological unsuitability or extreme claustrophobia.
* Pregnancy or unknown pregnancy status.
* Clinical instability as deemed by the attending physician; including but not limited to: cardiogenic shock, hypotension (systolic blood pressure < 90 mmHg), refractory hypertension (systolic blood pressure > 180 mmHg), sustained ventricular or atrial arrhythmia requiring intravenous medications.
* Use of Viagra or Cialis in the past 24 hours.
* Known history of allergy or adverse reactions to x-ray dye, regadenoson or aminophylline.
* Use of caffeine within the previous 12 hours (inactivates regadenoson).
* History of severe aortic stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients who have undergone a clinically indicated CCTA for suspicion of coronary artery disease and have a suspected coronary stenosis ≥50%-69% on that examination.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as a result of CTP procedure. | Through study completion, expected 1 year.
  Safety will be monitored by medical personnel and recorded from observations, patient interviews and the medical record during the index hospital visit(s) for CTP, from the medical record, and outpatient office records.

SECONDARY OUTCOMES:
Number of days for a subject to be scheduled and complete CTP procedure post CCTA procedure. | 30 days
  Days from CCTA to completed CTP procedure.
Number of minutes it takes for CTP procedure to be completed on a subject. to complete a CTP procedure. | 90 minutes
  Time (minutes) from initiation to completion of CTP procedure.
Number of minutes for a Provider to review and interpret CTP data and report out on CTP procedure. | 30 minutes
  Time (minutes) to interpret the CTP procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Jacob, MD, Principal Investigator — Lancaster General Health / Penn Medicine
Locations (1):
- Lancaster General Heatlh / Penn Medicine, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
An abstract reporting out on clinical study will be submitted for publication.
Supporting Information: CSR
Time Frame: April 2018
Access Criteria: Toshiba, Astellas

REFERENCES:
- [Background] Budoff MJ, Dowe D, Jollis JG, Gitter M, Sutherland J, Halamert E, Scherer M, Bellinger R, Martin A, Benton R, Delago A, Min JK. Diagnostic performance of 64-multidetector row coronary computed tomographic angiography for evaluation of coronary artery stenosis in individuals without known coronary artery disease: results from the prospective multicenter ACCURACY (Assessment by Coronary Computed Tomographic Angiography of Individuals Undergoing Invasive Coronary Angiography) trial. J Am Coll Cardiol. 2008 Nov 18;52(21):1724-32. doi: 10.1016/j.jacc.2008.07.031. PMID 19007693
- [Background] Hamon M, Biondi-Zoccai GG, Malagutti P, Agostoni P, Morello R, Valgimigli M, Hamon M. Diagnostic performance of multislice spiral computed tomography of coronary arteries as compared with conventional invasive coronary angiography: a meta-analysis. J Am Coll Cardiol. 2006 Nov 7;48(9):1896-910. doi: 10.1016/j.jacc.2006.08.028. Epub 2006 Sep 26. PMID 17084268
- [Background] Meijboom WB, Meijs MF, Schuijf JD, Cramer MJ, Mollet NR, van Mieghem CA, Nieman K, van Werkhoven JM, Pundziute G, Weustink AC, de Vos AM, Pugliese F, Rensing B, Jukema JW, Bax JJ, Prokop M, Doevendans PA, Hunink MG, Krestin GP, de Feyter PJ. Diagnostic accuracy of 64-slice computed tomography coronary angiography: a prospective, multicenter, multivendor study. J Am Coll Cardiol. 2008 Dec 16;52(25):2135-44. doi: 10.1016/j.jacc.2008.08.058. PMID 19095130
- [Background] Miller JM, Rochitte CE, Dewey M, Arbab-Zadeh A, Niinuma H, Gottlieb I, Paul N, Clouse ME, Shapiro EP, Hoe J, Lardo AC, Bush DE, de Roos A, Cox C, Brinker J, Lima JA. Diagnostic performance of coronary angiography by 64-row CT. N Engl J Med. 2008 Nov 27;359(22):2324-36. doi: 10.1056/NEJMoa0806576. PMID 19038879
- [Background] Abdulla J, Asferg C, Kofoed KF. Prognostic value of absence or presence of coronary artery disease determined by 64-slice computed tomography coronary angiography a systematic review and meta-analysis. Int J Cardiovasc Imaging. 2011 Mar;27(3):413-20. doi: 10.1007/s10554-010-9652-x. Epub 2010 Jun 12. PMID 20549366
- [Background] Gallagher MJ, Ross MA, Raff GL, Goldstein JA, O'Neill WW, O'Neil B. The diagnostic accuracy of 64-slice computed tomography coronary angiography compared with stress nuclear imaging in emergency department low-risk chest pain patients. Ann Emerg Med. 2007 Feb;49(2):125-36. doi: 10.1016/j.annemergmed.2006.06.043. Epub 2006 Sep 15. PMID 16978738
- [Background] Goldstein JA, Gallagher MJ, O'Neill WW, Ross MA, O'Neil BJ, Raff GL. A randomized controlled trial of multi-slice coronary computed tomography for evaluation of acute chest pain. J Am Coll Cardiol. 2007 Feb 27;49(8):863-71. doi: 10.1016/j.jacc.2006.08.064. Epub 2007 Feb 12. PMID 17320744
- [Background] Goldstein JA, Chinnaiyan KM, Abidov A, Achenbach S, Berman DS, Hayes SW, Hoffmann U, Lesser JR, Mikati IA, O'Neil BJ, Shaw LJ, Shen MY, Valeti US, Raff GL; CT-STAT Investigators. The CT-STAT (Coronary Computed Tomographic Angiography for Systematic Triage of Acute Chest Pain Patients to Treatment) trial. J Am Coll Cardiol. 2011 Sep 27;58(14):1414-22. doi: 10.1016/j.jacc.2011.03.068. PMID 21939822
- [Background] George RT, Arbab-Zadeh A, Cerci RJ, Vavere AL, Kitagawa K, Dewey M, Rochitte CE, Arai AE, Paul N, Rybicki FJ, Lardo AC, Clouse ME, Lima JA. Diagnostic performance of combined noninvasive coronary angiography and myocardial perfusion imaging using 320-MDCT: the CT angiography and perfusion methods of the CORE320 multicenter multinational diagnostic study. AJR Am J Roentgenol. 2011 Oct;197(4):829-37. doi: 10.2214/AJR.10.5689. PMID 21940569
- [Background] Rochitte CE, George RT, Chen MY, Arbab-Zadeh A, Dewey M, Miller JM, Niinuma H, Yoshioka K, Kitagawa K, Nakamori S, Laham R, Vavere AL, Cerci RJ, Mehra VC, Nomura C, Kofoed KF, Jinzaki M, Kuribayashi S, de Roos A, Laule M, Tan SY, Hoe J, Paul N, Rybicki FJ, Brinker JA, Arai AE, Cox C, Clouse ME, Di Carli MF, Lima JA. Computed tomography angiography and perfusion to assess coronary artery stenosis causing perfusion defects by single photon emission computed tomography: the CORE320 study. Eur Heart J. 2014 May;35(17):1120-30. doi: 10.1093/eurheartj/eht488. Epub 2013 Nov 19. PMID 24255127